CLINICAL TRIAL: NCT03856801
Title: Acute Effects of Whole-body Vibration Training in Hypoxia and Normoxia Condition on Neuromuscular Performance and Mobility in Patients With Multiple Sclerosis
Brief Title: Acute Effects of Whole-body Vibration Training in Hypoxia and Normoxia in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio, Profesor Titular, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE061908
Record Dates: First submitted 2019-02-13; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Multiple Sclerosis
Keywords: neuromuscular disease; whole-body vibration; hypoxia; strength
MeSH Terms: conditions — Multiple Sclerosis; Neuromuscular Diseases; Hypoxia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body vibration in normoxia condition (Experimental): Training session in normoxia condition
  Interventions: Other: Exercise
- Whole-body vibration in hypoxia condition (Experimental): Training session in hypoxia condition
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Whole-body vibration training in hypoxia and normoxia condition

SUMMARY:
Multiple Sclerosis (ME) is a degenerative, inflammatory and autoimmune demyelinating disease of the central nervous system, characterized by demyelination due to inflammation and degeneration of the myelin sheaths enveloping nerves of the eye, periventricular grey matter, brain, spinal cord and brainstem. The symptoms associated with MS include symptomatic fatigue, muscle weakness, ataxia, mobility and balance problems or cognitive problems. Moderate intensity strength training has been shown to improve strength and mobility in persons with MS. It was suggested that whole-body vibration training (WBVT) is effective to improve muscle strength, such as resistance training, resulting from both neural and structural adaptations. On the other hand, traditional strength training in hypoxia has garnered much attention. This method has shown improvements in isometric strength and increases in muscle size.

DETAILED DESCRIPTION:
* Crossover.
* 13 patients with multiple sclerosis were recruited.
* Patients performed two sessions: whole-body vibration training in normoxia condition and whole-body vibration in hypoxia condition.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate disability with clinical mild spastic-ataxic gait disorder.
* stable phase of the disease.

Exclusion Criteria:

* Expanded Disability Status Scale (EDSS) < 6.
* relapsing disease within the preceding 12 months.
* corticosteroid treatment within the last months before study inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction of Knee Extension | Immediately before the training sessions
Maximal Voluntary Isometric Contraction of Knee Extension | Immediately after the training sessions
Rate of Force Development | Immediately before the training sessions
Rate of Force Development | Immediately after the training sessions
Central Activation Ratio | Immediately before the training sessions
Central Activation Ratio | Immediately after the training sessions
Biomechanical study of the walk by video recording | Immediately before the training sessions
  Kinematic analysis of knee and ankle angles during walking
Biomechanical study of the walk by video recording | Immediately after the training sessions
  Kinematic analysis of knee and ankle angles during walking
Biomechanical study of the walk by video recording | Immediately before the training sessions
  Stride amplitude during walking
Biomechanical study of the walk by video recording | Immediately after the training sessions
  Stride amplitude during walking
Spasticity | Immediately before the training sessions
  Pendulum test
Spasticity | Immediately after the training sessions
  Pendulum test

SECONDARY OUTCOMES:
Rate of Perceived Exertion | Immediately before the training sessions
  RPE Scale 6-20
Rate of Perceived Exertion | Immediately after the training sessions
  RPE Scale 6-20
Walking speed | Immediately before the training sessions
  Test 10 m-walks
Walking speed | Immediately after the training sessions
  Test 10 m-walks
Static balance | Immediately before the training sessions
  Romberg Test with eyes open and closed. Analysis with force plates
Static balance | Immediately after the training sessions
  Romberg Test with eyes open and closed. Analysis with force plates
Muscle oxygenation in soleus | Immediately before the training sessions
  MOXY's
Muscle oxygenation in soleus | Immediately after the training sessions
  MOXY's

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided